CLINICAL TRIAL: NCT03979235
Title: Developing Clinic-oriented Quantitative Effectiveness Evaluation and Individualized Therapeutic Programs of Rehabilitation
Brief Title: Developing Effectiveness Evaluation and Therapeutic Programs of Rehabilitation
Status: Recruiting | Type: Observational
Sponsor: National Research Center for Rehabilitation Technical Aids (Other)
Responsible Party: Principal Investigator, Pengxu Wei, Director, National Research Center for Rehabilitation Technical Aids
Other Study IDs: 20180104
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers; Motor Deficits; Dysphagia
MeSH Terms: conditions — Neurologic Manifestations; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heahlthy people: perform motor function assessment by using scales, sEMG, and inertia sensors
  Interventions: Diagnostic Test: Motor function assessment
- People with motor deficits: perform motor function assessment by using scales, sEMG, and inertia sensors
  Interventions: Diagnostic Test: Motor function assessment
- Patients with dysphagia: perform motor function assessment by using scales, sEMG, and inertia sensors
  Interventions: Diagnostic Test: Motor function assessment

INTERVENTIONS:
Diagnostic Test: Motor function assessment — perform motor function assessment by using scales, sEMG, and inertia sensors

SUMMARY:
Using robotics, sensors, and sEMG to develop clinic-oriented quantitative effectiveness evaluation and individualized programs of rehabilitation

DETAILED DESCRIPTION:
Using robotics, sensors, sEMG or other methods to develop clinic-oriented quantitative effectiveness evaluation and individualized programs of rehabilitation

ELIGIBILITY:
Inclusion Criteria (for healthy people):

* no history of psychological/psychotic problems, no history of important diseases.

Exclusion Criteria (for healthy people):

* history of psychological/psychotic problems

Inclusion Criteria (for patients with motor deficits or dysphagia):

* patients with motor function impairment such as post stroke hemiplegia.

Exclusion Criteria (for patients with motor deficits or dysphagia):

* cognitively or physically unable to cooperate with the examiner to finish the test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruiting with advertising
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-06-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor function assessment | Change from Baseline scores at 1 month
  Fugl-Meyer Assessment

SECONDARY OUTCOMES:
surface EMG | Change from Baseline status at 1 month
  high-density surface EMG
Kinematics test | Change from Baseline status at 1 month
  Using inertia sensors to assess kinematics during movement

CONTACTS AND LOCATIONS:
Overall Officials: PX Wei, PhD, Principal Investigator — National Research Center for Rehabilitation Technical Aids
Locations (1):
- National Research Center for Rehabilitation Technical Aids, Beijing, China